CLINICAL TRIAL: NCT00646880
Title: Double-Blind Crossover Comparative Ambulatory Urodynamic Monitoring (AUM) Study of Tolterodine PR and Propiverine in Korean Patients With Overactive Bladder (OAB)
Brief Title: A Study to Evaluate the Efficacy of Tolterodine Prolonged Release Compared With Propiverine for the Treatment of Korean Patients With Overactive Bladder as Assessed by Ambulatory Urodynamic Monitoring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DETAOD-0084-055
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Urinary Bladder, Overactive
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — propiverine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Propiverine/tolterodine group (Active Comparator)
  Interventions: Drug: propiverine
- Tolerodine/propiverine group (Active Comparator)
  Interventions: Drug: tolterodine PR

INTERVENTIONS:
Drug: propiverine — Two week washout period followed by propiverine 20 mg capsule daily for 1 week, followed by a second 2-week washout; patients were then crossed over to tolterodine PR 4 mg capsule daily for 1 week.
  Arms: Propiverine/tolterodine group
Drug: tolterodine PR — Two week washout period followed by tolterodine PR 4 mg capsule daily for 1 week, followed by a second 2-week washout; patients were then crossed over to propiverine 20 mg capsule daily for 1 week.
  Arms: Tolerodine/propiverine group

SUMMARY:
The purpose of this study is to compare the difference between tolterodine prolonged release (PR) and propiverine in efficacy as assessed by the AUM and to show that tolterodine PR is similar to propiverine with respect to micturition chart variables and safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of urinary urgency
* Symptoms of urinary frequency (greater than or equal to 8 micturitions per 24 hours) as verified on the patient's micturition chart
* Symptoms of overactive bladder for greater than or equal to 6 months

Exclusion Criteria:

* Stress incontinence as determined by the investigator and confirmed for female patients by a cough provocation test
* An average volume voided of >200 ml per micturition as verified on the micturition chart before randomization
* Total daily urine volume of >3000 ml as verified on the micturition chart before randomization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-03; Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Parameters of detrusor activity, occurring throughout the duration of comparable AUM | 28 days

SECONDARY OUTCOMES:
Number of pads used per 24 hours | 28 days
Urge Incontinence | 28 days
Number of urgency episodes | 28 days
Number of micturitions per 24 hours | 28 days
Volume voided per micturition | 28 days
Patient's perception of bladder condition | 28 days
Patient's perception of treatment benefit | 28 days
Patient's perception of urgency | 28 days
The occurrences of adverse events and withdrawals and changes in laboratory variables over each 1-week treatment period. | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=DETAOD-0084-055&StudyName=A%20Study%20to%20Evaluate%20the%20Efficacy%20of%20Tolterodine%20Prolonged%20Release%20Compared%20with%20Propiverine%20for%20the%20Treatment%20of%20Korean%20Patients%20